CLINICAL TRIAL: NCT07023926
Title: The Efficacy and Safety of Acupuncture for Prophylaxis of Menstrually Related Migraine: a Pilot Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Acupuncture for Prophylaxis of Menstrually Related Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, weiming wang, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-031-KY-01
Record Dates: First submitted 2025-05-29; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Menstrually Related Migraine; Electroacupuncture
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elecrtoacupuncture group (EA group) (Experimental): Participants will be treated by electroacupuncture. During the first week (from day -3 to +4 of menstruation), they will receive 1-2 sessions, followed by 2-3 sessions per week for the next three weeks. This treatment schedule will be repeated for three consecutive menstrual cycles, totaling a 12-week treatment period and 30 sessions. All treatment sessions will be monitored and recorded using a treatment diary.
  Interventions: Device: electroacupuncture
- Sham elecrtoacupuncture group (sham EA group) (Sham Comparator): Participants will be treated by sham electroacupuncture. The treatment frequency and sessions will be the same as in EA group, and the treatment diary will also be used in SEA group.
  Interventions: Device: Sham electroacupuncture

INTERVENTIONS:
Device: electroacupuncture — The supine position, the local skin of the acupoints was routinely sterilized, and the selected acupoints were pasted with Acupuncture auxiliary device. The main acupuncture points are DU20, bilateral EX-HN5, ST8, GB20, GB20, LI4, LR3, ST40. Select compatible acupoints based on the patient's accompanying symptoms: 1.Discomfort in the neck: EX-B2 of Cervical 3-4; 2.Emotional anxiety, depression or sleep disorders: GV29, HT7; 3.Stomach or abdominal discomfort: CV12, ST25 and CV6. The disposable acupuncture needles and the electronic acupuncture treatment instrument SDZ-V nerve and muscle intimulator both manufactured by Suzhou Medical Appliance Factory Co., Ltd., China.The specifications of acupuncture needles are Φ0.30×25mm, Φ0.30×40mm. The needles will be inserted into the skin of acupuncture points and manipulated manually by using the techniques such as lifting, thrusting, and twirling, until the internal compound sensation known as deqi.
  Arms: elecrtoacupuncture group (EA group)
Device: Sham electroacupuncture — The SEA group will use Hua Tuo brand disposable blunt-tip sham needles (Φ0.3mm×25mm) and the electronic acupuncture treatment instrument SDZ-V nerve and muscle intimulator both manufactured by Suzhou Medical Appliance Factory Co., Ltd., China. Sham points 1-2, 3-4, 5-6, and 7-8 are bilaterally located at the midpoints between the following pairs of acupoints: SP19 and EX-UE12, SP6 and LR5, EX-UE1 and HT1, and HT7 and SI8. sham LI4: Bilateral of midpoint between acupoint LI4 and LU9; sham LR3: Bilateral of midpoint between acupoint LR3 and ST44; sham ST40: Bilateral of midpoint between acupoint ST40 and GB35. Compatible acupoints: EX-B2 of Cervical 3-4 horizontal side by 0.5 cun; sham GV29: midpoint between acupoint GV29 and BL2. sham CV12: midpoint between acupoint CV12 and ST21; sham ST25: Bilateral of midpoint between acupoint ST25 and SP15; sham CV6: 3 cun lateral to the level of the CV6; The width of the interphalangeal joint of the patient's thumb was 1 "cun".
  Arms: Sham elecrtoacupuncture group (sham EA group)

SUMMARY:
Acupuncture is commonly used for the prevention of migraine and tension-type headaches, and has been found to be effective in reducing both the frequency and severity of these conditions. However, studies on acupuncture for menstrually related migraine (MRM) are limited, and current research has not been able to determine whether its efficacy is due to the actual therapeutic effects of acupuncture or psychological benefits. To address this issue, the investigators have designed a clinical trial to evaluate the efficacy of acupuncture for MRM.

ELIGIBILITY:
Inclusion Criteria:

1. meet the diagnostic criteria for MRM according to the ICHD-3, with a documented history of MRM for at least 12 months;
2. have a confirmed diagnosis of migraine by a neurologist;
3. aged 18-45 years;
4. have regular menstrual cycles (28 ± 7 days) with menstruation lasting 3-7 days;
5. have experienced ≥3 headache days during each menstrual cycle (days -2 to +3) and ≥5 total headache days per cycle over the past 3 months and baseline period; migraine attacks must last 4-72 hours without acute medication, or at least 2 hours when treated;
6. have completed a headache diary during the screening period (covering at least one full menstrual cycle), demonstrating good compliance;
7. headache diary data during screening period must meet the ICHD-3 criteria for MRM and fulfill criteria (4) and (5);
8. voluntarily sign the informed consent.

Exclusion Criteria:

1. irregular menstrual cycles, defined as cycle length outside the range of 28±7 days or menstruation duration <3 days or >7 days;
2. presence of secondary headache disorders, facial neuralgia, or cranial neuralgia;
3. combined with serious primary diseases such as cardiovascular, hepatic, renal, gastrointestinal, or hematological disorders that may interfere with the treatment protocol, or comorbid neurological conditions such as epilepsy, parkinson's disease, or other central nervous system disorders;
4. headache symptoms caused by other conditions, such as moderate to severe head or neck trauma, perimenstrual infections, intracranial tumors, intracranial infections, endocrine or metabolic disorders;
5. receipt of preventive treatment for headache within 1 month prior to the screening visit;
6. afraid of needles or received acupuncture treatment within 3 months;
7. unwillingness to undergo the study intervention or failure to sign the informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in standardized monthly headache days (SMHD) compared with baseline. | At Week 12 post-treatment
  The primary outcome is the change in standardized monthly headache days (SMHD). SMHD are calculated by adjusting the actual number of headache days to a standard 28-day menstrual cycle using the following formula: SMHD = (actual headache days × 28) ÷ individual menstrual cycle length

SECONDARY OUTCOMES:
change in standardized monthly headache days (SMHD) compared with baseline | At Weeks 4 and 8 post-treatment, and at Weeks 16, 20, and 24 during follow-up
The proportion of patients with cured MRM | At Week 12 post-treatment, and at weeks 16, 20, and 24 during follow-up
  Patients are defined as cured if they no longer met the diagnostic criteria for MRM.
The responder rate | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  The responder rate is defined as a minimum of 50 % reduction in SMHD compared with baseline.
Change in standardized monthly headache severity score from baseline | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  Standardized monthly headache severity score = (Actual monthly severity score × 28) ÷ Individual menstrual cycle length.
Change in standardized monthly use of rescue medication from baseline | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  Rescue medication taken standardized monthly = (Actual doses × 28) ÷ Individual menstrual cycle length
Headache diary completion rate | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  Headache diary completion rate
Overall recruitment rate at End of recruitment phase | At end of the recruitment phase
  Recruitment rate = (Number of enrolled participants ÷ Total number of eligible patients) × 100%.
Overall retention rate | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  Retention rate = (Number of participants who completed the study ÷ Total enrolled participants) × 100%.
Change in Hospital Anxiety and Depression Scale (HADS) score from baseline | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  The HADS is a validated self-report questionnaire used to assess symptoms of anxiety and depression over the past week. It consists of 14 items divided into two subscales: anxiety and depression, each containing 7 items. Each item is rated on a 4-point scale (0-3), yielding subscale scores ranging from 0 to 21. Higher scores reflect greater symptom severity.
Change in Headache Impact Test-6 (HIT-6) score from baseline | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  The HIT-6 is a validated, self-reported instrument used to assess the impact of headaches on health-related quality of life. It includes six items covering domains such as pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. Each item is scored on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The total score ranges from 36 to 78, with higher scores indicating greater headache-related disability.
Change in Migraine-Specific Quality of Life Questionnaire (MSQ v2.1) score from baseline | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  The MSQ v2.1 assesses migraine-related quality of life across three domains: Role Function-Restrictive , Role Function-Preventive , and Emotional Function. Each item is rated on a 6-point Likert scale from 1 ("All the time") to 6 ("None of the time"). Domain scores are calculated and transformed to a 0-100 scale, with higher scores indicating better quality of life.
Patient's Global Impression of Change (PGIC) | At Weeks 4, 8, and 12 post-treatment, and at Weeks 16, 20, and 24 during follow-up
  The PGIC scale will be used to assess participants' subjective perception of overall improvement. It is a 7-point scale with the following categories: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Lower scores indicate greater perceived improvement.
Participants' expectation for acupuncture | At baseline
  Participants will be asked the following question to assess their expectations regarding acupuncture for MRM: "What level of improvement do you expect from acupuncture for your MRM?" Response options will include: "no improvement," "slight improvement," "moderate improvement," "marked improvement," and "unclear." The association between participants' expectations and the primary outcome will be examined using statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Wang, Ph.D, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Department of Acupuncture, China Academy of Chinese Medical Sciences Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available on reasonable request. You can send e-mail to us if you have any question
Supporting Information: Study Protocol, SAP
Time Frame: It depends
Access Criteria: It depends

REFERENCES:
- [Derived] Liu X, Jiao R, Zheng Y, Liu Y, Yu G, Shi J, Wang W, Wang W. The Efficacy and Safety of Electroacupuncture for Prophylaxis of Menstrually Related Migraine: Study Protocol for a Pilot Randomized Controlled Trial. Int J Womens Health. 2025 Oct 8;17:3541-3555. doi: 10.2147/IJWH.S548053. eCollection 2025. PMID 41084597